CLINICAL TRIAL: NCT00445627
Title: Natural History of Type 2 Diabetes Mellitus in Children and Young Adults
Brief Title: Effect of Short-Term Beta-Cell Rest in Adolescents and Young Adults With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070115; 07-DK-0115
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01-27

CONDITIONS: Obesity; Overweight; Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Obesity; Insulin; Metformin; Natural History; Overweight
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Metformin; Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Lean Controls: Cross-sectional analyses of continuous variables (e.g. hormonal measurements, inflammatory markers, lipids, BMI, and body composition measurements) will be compared using ANOVA
  Interventions: Behavioral: Nutrition counseling; Behavioral: Exercise counseling
- Overweight Obese Controls: Cross-sectional analyses of continuous variables (e.g. hormonal measurements, inflammatory markers, lipids, BMI, and body composition measurements) will be compared using ANOVA
  Interventions: Drug: Metformin; Behavioral: Nutrition counseling; Behavioral: Exercise counseling
- Type 1 Diabetes: Cross-sectional analyses of continuous variables (e.g. hormonal measurements, inflammatory markers, lipids, BMI, and body composition measurements) will be compared using ANOVA
  Interventions: Drug: Insulin; Behavioral: Nutrition counseling; Behavioral: Exercise counseling

INTERVENTIONS:
Drug: Metformin
  Groups: Overweight Obese Controls
Drug: Insulin
  Groups: Type 1 Diabetes
Behavioral: Nutrition counseling
Behavioral: Exercise counseling

SUMMARY:
This study will determine whether resting beta cells (cells in the pancreas that produce insulin) for 2 weeks will improve the ability of patients with Type 2 diabetes mellitus (T2DM) to make insulin. Beta cells can rest by giving patients insulin shots. The study will also examine how teenagers with T2DM feel about having diabetes and explore differences between young people with and without T2DM.

This study includes patients 12 to 25 years of age with T2DM who are overweight and who were diagnosed within 2 years of enrolling in the study. Healthy individuals of normal weight or who are overweight are also eligible. Candidates are screened with a medical history, physical examination and laboratory tests.

Participants with T2DM are assigned to one of two groups. Group 1 takes an anti-diabetes medicine called metformin and follows a diet prescribed by a study staff dietitian for 2 weeks. Group 2 takes metformin, follows the prescribed diet, and receives insulin through a pump under the skin for 2 weeks. During these two weeks, all participants have the following tests:

* Frequent blood sugar checks.
* Oral glucose tolerance test (routine diabetes test in which blood samples are drawn before and several times after the subject drinks a sugary solution).
* Arginine stimulation to test the response of the body to arginine, a normal ingredient of food that stimulates the release of insulin. Two catheters are placed into veins in the arms, one to administer a liquid containing arginine, the other to draw the blood samples.
* Ultrasound of the blood vessels in the neck to check for hardening of the arteries.
* Metabolism test to measure the amount of oxygen used during rest. The subject breathes normally during rest while wearing a canopy over his or her head for about 20 minutes.
* MRI scans of the abdomen to examine the amount of fat in the belly (at the beginning and end of the study)
* DEXA scan to determine percent body fat.
* Tests to explore quality of life and feelings about health, work or school, friends and family.
* Exercise testing on a treadmill or stationary bicycle.
* Genetic studies for information on diabetes and obesity.

Normal volunteers have blood draws, oral glucose tolerance testing, MRI scan, DEXA scan, psychological testing, exercise testing, and genetic testing.

DETAILED DESCRIPTION:
Background:

Type 2 diabetes mellitus (T2DM) is a condition characterized by insulin resistance and progressive failure of the insulin-secreting beta-cells. Previously considered a disease of adults, it is now becoming increasingly prevalent in children and adolescents. Patients with childhood onset T2DM are at very high risk for diabetes-related morbidity and mortality, due to a longer life-time duration of diabetes, as well as possible increased rapidity of Beta-cell failure.

Aims:

In this study, we will address the following aims:

1. To characterize hormonal, metabolic, and behavioral traits in patients with youth-onset type 2 diabetes. These will include:

   1. Assessment of Beta-cell function and insulin resistance
   2. Psychological, demographic, and socioeconomic assessments
   3. Assessment of the physiology and pathophysiology of incretins and other gut hormones
   4. Identification of early biomarkers of diabetes complications, especially cardiovascular disease
   5. Validation of new methods for studying glucose metabolism
2. To serve as a recruitment and development tool for hypothesis-driven pilot studies, discussed in the appendices of this protocol.

Methods:

Children and young adults ages 8 to 25 years with type 2 diabetes will be studied in a cross-sectional and longitudinal manner. Two control groups without diabetes will be studied for comparison purposes: healthy lean controls, and overweight/obese controls. Methods used to study participants include routine blood sampling, oral glucose tolerance testing, mixed meal testing, arginine stimulation testing, DEXA, MRI, carotid ultrasound, questionnaires, exercise physiology, and measurements of energy expenditure. Patients with type 1 diabetes will be studied using oral glucose tolerance and mixed meal tests in a pilot study of artificial sweeteners.

ELIGIBILITY:
* DIABETIC SUBJECTS:

INCLUSION CRITERIA:

1. Type 2 diabetes mellitus as defined by:

   1. Fasting blood glucose greater than or equal to 126 mg/dL OR postprandial blood sugar greater than or equal to 200 mg/dL (either during OGTT at NIH or as previously documented on outside medical record).
   2. Since subjects may already have been started on treatment with hypoglycemic agents at the time of enrollment, they may have blood glucose levels in the impaired glucose tolerance range (fasting glucose 100-125 mg/dL and postprandial 140-199 mg/dL). This is a sign of adequately controlled diabetes, rather than an incorrect diagnosis of diabetes. Therefore, prior documentation (on outside medical records) of blood glucose values documenting diabetes will be acceptable if the subject has impaired glucose tolerance rather than overt diabetes according to screening results at NIH.
   3. Absence of insulin autoantibodies (in insulin na(SqrRoot) ve patients only)

   Or
2. Clinical diagnosis of type 1 diabetes mellitus (for Pilot Study only)

   And
3. Age 8-25 years at enrollment

EXCLUSION CRITERIA:

1. Normal OGTT at NIH (fasting blood glucose < 100 mg/dL AND 2 hour blood glucose < 140 mg/dL)
2. Significant comorbidity that, in the opinion of the investigators, will increase risk to the subject(specific obesity-related comorbidities are explicitly permitted, including hypertension, hyperlipidemia, obstructive sleep apnea and non-alcoholic steatohepatitis)
3. Positive urine pregnancy test
4. Psychiatric or cognitive disorder that will, in the opinion of the investigators, limit the subject's ability to comply with study procedures

NON-DIABETIC CONTROLS:

INCLUSION CRITERIA:

Two types of volunteers will be recruited:

1. Overweight and obese volunteers who will be BMI matched with study enrollees who have T2DM during analyses
2. Normal weight (BMI between 5th and 85th centiles for age) volunteers

EXCLUSION CRITERIA:

1. Diabetes
2. Significant comorbidity that, in the opinion of the investigators, will increase risk to the subject (specific obesity-related comorbidities are explicitly permitted, including hypertension, hyperlipidemia, obstructive sleep apnea and non-alcoholic steatohepatitis)
3. Current use of drugs that alter glucose metabolism (e.g. metformin)
4. Current use of prescription or non-prescription weight-loss drugs
5. Positive urine pregnancy test
6. Psychiatric or cognitive disorder that will, in the opinion of the investigators, limit the subject's ability to comply with study procedures

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults ages 8 to 25 years with type 2 diabetes will be studied in a cross-sectional and longitudinal manner.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-06-18 (Actual)

PRIMARY OUTCOMES:
evaluate phenotype of T2DM | 20 months
  Measurements will include indices of beta-cell function, body composition, cardiovascular disease risk factors, gut hormones, and psychological well-being. These data will be compared to findings in non-diabetic volunteers who are lean or overweight/obese

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Chung, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dabelea D, Hanson RL, Bennett PH, Roumain J, Knowler WC, Pettitt DJ. Increasing prevalence of Type II diabetes in American Indian children. Diabetologia. 1998 Aug;41(8):904-10. doi: 10.1007/s001250051006. PMID 9726592
- [Background] Fridlyand LE, Philipson LH. Does the glucose-dependent insulin secretion mechanism itself cause oxidative stress in pancreatic beta-cells? Diabetes. 2004 Aug;53(8):1942-8. doi: 10.2337/diabetes.53.8.1942. PMID 15277370
- [Background] Gungor N, Bacha F, Saad R, Janosky J, Arslanian S. Youth type 2 diabetes: insulin resistance, beta-cell failure, or both? Diabetes Care. 2005 Mar;28(3):638-44. doi: 10.2337/diacare.28.3.638. PMID 15735201
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-DK-0115.html